CLINICAL TRIAL: NCT02531906
Title: Analysis of Analgesia Regimens During Concurrent Chemoradiation for Head and Neck Cancer: A Pilot Study
Brief Title: Gabapentin, Methadone Hydrochloride, and Oxycodone Hydrochloride in Improving Quality of Life in Patients With Stage II-IV Head and Neck Cancer During Chemoradiation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 262314; NCI-2015-01338 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 262314 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2015-08-19; First posted 2015-08-25 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Pain; Stomatitis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Pain; Stomatitis | interventions — Gabapentin; Methadone; Amidines; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (gabapentin) (Experimental): Patients receive gabapentin PO TID for up to 7 weeks during radiotherapy.
  All patients may continue to receive treatment for pain throughout their course of chemoradiation therapy (and up to 24 months following CRT if continuing on a pain regimen).
  Interventions: Drug: Gabapentin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (gabapentin, methadone, oxycodone) (Experimental): Patients receive gabapentin PO TID, methadone hydrochloride PO BID, and oxycodone hydrochloride PO Q8H PRN for up to 7 weeks during radiotherapy.
  All patients may continue to receive treatment for pain throughout their course of chemoradiation therapy (and up to 24 months following CRT if continuing on a pain regimen).
  Interventions: Drug: Gabapentin; Drug: Methadone Hydrochloride; Drug: Oxycodone Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Gabapentin — Given PO
  Other Names: Gralise; Neurontin
Drug: Methadone Hydrochloride — Given PO
  Other Names: Adanon; Althose; Dolophine; Methadose
  Arms: Arm II (gabapentin, methadone, oxycodone)
Drug: Oxycodone Hydrochloride — Given PO
  Other Names: Oxecta; OxyContin; Roxicodone
  Arms: Arm II (gabapentin, methadone, oxycodone)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the side effects of gabapentin and how well it works when given together with methadone hydrochloride and oxycodone hydrochloride in improving quality of life in patients with stage II-IV head and neck cancer during chemoradiation. Gabapentin, methadone hydrochloride, and oxycodone hydrochloride may help relieve moderate or severe pain caused by head and neck cancer during and after chemoradiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Collect preliminary data on the safety and efficacy of two analgesic regimens that can be used to design larger studies for comparing such regimens.

SECONDARY OBJECTIVES:

I. Examine effects of the treatment regimens on pain control, oral mucositis, and quality-of-life ratings scores during and after chemoradiation therapy (CRT).

TERTIARY OBJECTIVES:

I. To assess treatment regimen effect on patient nutrition and hydration status during and after CRT (weight loss, vitals, oral [PO] tolerance, etc.).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive gabapentin PO thrice daily (TID) for up to 7 weeks during radiotherapy.

ARM II: Patients receive gabapentin PO TID, methadone hydrochloride PO twice daily (BID), and oxycodone hydrochloride PO every 8 hours (Q8H) as needed (PRN) for up to 7 weeks during radiotherapy.

All patients may continue to receive treatment for pain throughout their course of chemoradiation therapy (and up to 24 months following CRT if continuing on a pain regimen).

After completion of study, patients are followed up at 30 days, and at 3, 6, 9, and 12 months. Patients requiring prolonged analgesic therapy may be followed up every 6 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for chemoradiation therapy of the head and neck
* Baseline creatinine (Cr) no greater than 1.5 times the upper limit of normal
* Have a clinical stage II-IV head and neck carcinoma
* Have a pathologic diagnosis of squamous cell carcinoma of the head and neck region
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Ability to swallow and retain oral medication or take through a feeding tube
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have previously been treated with surgery or radiation for head and neck cancer and/or are being treated for recurrent head and neck cancer
* Patients with known brain metastases will be excluded from this clinical trial
* Any patients prescribed medications for chronic pain and/or neuropathy will be excluded, including patients under treatment of a pain specialist or substance-abuse programs
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Patients on medications that prolong QT interval
* Patients on dialysis or with transplanted organs
* Patients already enrolled on other studies of systemic pain control agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-24; Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Change in pain levels via Oral Mucositis Daily Questionnaire (OMDQ), European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30, Head and Neck Quality of Life Survey, and physical evaluations | Baseline to up to 24 months
  Evaluated using a repeated measures model. Tested using a two-sided 0.05 significance level. Post hoc analyses will be done with multiple comparisons adjusted for using the Bonferroni method. Assumptions of normality and equal variance will be examined, and transformations will be used as appropriate.
Incidence of side effects or drug intolerance | Up to 24 months
  Will be graded and recorded. Tested using a two-sided 0.05 significance level. Post hoc analyses will be done with multiple comparisons adjusted for using the Bonferroni method. Assumptions of normality and equal variance will be examined, and transformations will be used as appropriate. The frequency of toxicities will be tabulated by grade by treatment arm.
Proportion of patients who require higher equivalents of narcotic support added to their analgesia regimen in each arm | Up to 24 months
  Each patient requiring rescue medication for breakthrough or refractory pain will be counted as a failure for that specific regimen. At the end of the trial, number of failures will be compared between the two treatment arms using Fisher's exact test. Total amount of opioid intake mean will be compared using a t-test between the two arms. Tested using a two-sided 0.05 significance level. Post hoc analyses will be done with multiple comparisons adjusted for using the Bonferroni method. Assumptions of normality and equal variance will be examined, and transformations will be used as appropriate

SECONDARY OUTCOMES:
Change in oral mucositis rating scores during and after CRT, using the OMDQ | Baseline to up to 24 months
  The total score of the OMDQ questionnaire will be recorded after each follow-up visit. Tested using a two-sided 0.05 significance level. Post hoc analyses will be done with multiple comparisons adjusted for using the Bonferroni method. Assumptions of normality and equal variance will be examined, and transformations will be used as appropriate.
Change in quality of life rating scores during and after CRT, using the EORTC QLQ-C30 and H&N35 | Baseline to up to 24 months
  The total score of the EORTC questionnaires will be recorded after each follow-up visit. Tested using a two-sided 0.05 significance level. Post hoc analyses will be done with multiple comparisons adjusted for using the Bonferroni method. Assumptions of normality and equal variance will be examined, and transformations will be used as appropriate.

OTHER OUTCOMES:
Change in patient hydration and nutrition using the OMDQ | Baseline to up to 24 months
  Tested using a two-sided 0.05 significance level. Post hoc analyses will be done with multiple comparisons adjusted for using the Bonferroni method. Assumptions of normality and equal variance will be examined, and transformations will be used as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States